CLINICAL TRIAL: NCT03708471
Title: Efficacy of Two-stage Hybrid Ablation or Thoracoscopic Epicardial Ablation for Long-standing Persistent Atrial Fibrillation: A Prospective, Randomized Controlled Trial
Brief Title: Two-stage Hybrid Ablation or Thoracoscopic Epicardial Ablation for Long-standing Persistent Atrial Fibrillation
Acronym: THAT-LSPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Huiming Guo, Director of department of adult cardiac surgery, Guangdong Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THAT-LSPAF
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Hybrid ablation; Surgical ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two-stage hybrid abltaion (Experimental): After thoracoscopic surgical ablation and 3 months of blanking-period, patients in this group will receive percutaneous catheter ablation and recommendations about cardiovascular risk control.
  Interventions: Procedure: Hybrid ablation
- Thoracosopic surgical ablation (Active Comparator): After thoracoscopic surgical ablation and 3 months of blanking-period, patients in this group will only receive recommendations about cardiovascular risk control.
  Interventions: Procedure: Thoracoscopic surgical ablation

INTERVENTIONS:
Procedure: Hybrid ablation — This intervention including thoracoscopic surgical ablation, percutaneous catheter ablation and cardiovascular risk control.
  Arms: Two-stage hybrid abltaion
Procedure: Thoracoscopic surgical ablation — This intervention including thoracoscopic surgical ablation and cardiovascular risk control.
  Arms: Thoracosopic surgical ablation

SUMMARY:
Hybrid ablation, as an emerging strategy for atrial fibrillation (AF) in recent years, shows encouraging outcomes in many medical centers. A lot of cases demonstrated hybrid ablation has higher success rate than surgical ablation on patients with persistent AF, especially long-standing persistent AF (LSPAF). But it is still lack of high level evidence to prove it.

This study focus on patients with long-standing persistent atrial fibrillation (LSPAF). In order to compare the efficacy and safety of hybrid ablation (two-stage) versus thoracoscopic surgical ablation, a randomized, controlled clinical trial will be performed in the population of LSPAF patients.

DETAILED DESCRIPTION:
In this study, all selected LSPAF patients will receive thoracoscopic surgical ablation. After 3 months of blanking-period, patients off antiarrhythmic therapy freedom from atrial arrhythmia (including atrial tachycardia, atrial flutter and atrial fibrillation) will be divided into Hybrid group and Surgical group randomly and equally. Patients of Hybrid group will receive transcatheter endocardial electrophysiological mapping and catheter ablation after randomization subsequently. In followed 2 years, cardiovascular risk control will be recommended to 2 groups' patients.

During the 2-year follow-up, 7d-Holter will be used to monitor patients' rhythm and cardiac conditions will be confirmed by transthoracic echocardiography (TTE). Physical examination and examinations mentioned above will be performed in 3 months, 6 months, 12 months, 18 months, 24 months and suspected recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Nonvalvular and long-standing persistent atrial fibrillation confirmed by echocardiography and electrocardiography respectively.
* Written informed consent

Exclusion Criteria:

* Secondary atrial fibrillation caused by other reversible diseases.
* Left atrial diameter >55mm confrimed by Transthoracic echocardiography.
* Intracardial mass or thrombus.
* Previous cardiac surgery.
* Uncontrolled heart failure or LVEF less than 30%.
* Severe chest wall deformity.
* Possibly pleural adhesion or pericardial adhesion caused by previous thoracic surgery, tuberculosis or constrictive pericarditis.
* Severe comorbidities (e.g. severe CAD, severe renal failure, severe liver failure).
* Life expectancy less than 2 years (e.g. patients with MODS or cancer)
* Unsuitable for radiation exposure (e.g. pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-03-04 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia recurrence | 24 months after blanking-period.
  Atrial arrhythmia (including atrial tachycardia, atrial flutter and atrial fibrillation) longer than 30s, off antiarrhythmic therapy, recorded by ECG or Holter.

SECONDARY OUTCOMES:
Systemic atrial embolism | 24 months after blanking-period.
  Including cerebral infarction and other peripheral atrial embolism
Left atrial thrombus | At 3months, 6months, 12months, 18months, 24months after intervention.
  New-onset left atrial thrombus confirmed by TEE or TTE

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China